CLINICAL TRIAL: NCT05427305
Title: Bevacizumab Biosimilar Candidate TAB008 Compared to Avastin® in Patients With Locally Advanced, Metastatic EGFR Wild-type Non-squamous Non-small Cell Lung Cancer: a Randomized, Double-blind, Multicenter Study
Brief Title: TAB008 Compared to Avastin® in Patients With EGFR Wild-type Non-squamous Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioDlink Biopharm Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TOT-CR-TAB008-Ⅲ-01
Record Dates: First submitted 2022-06-09; First posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Efficacy
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAB008 (Experimental): Eligible patients received TAB008 15 mg/kg every three weeks for 6 cycles, then 7.5mg/kg until disease progression, intolerable toxicity, withdrawal of consent, lost to follow up or death.
  Interventions: Drug: TAB008
- Bevacizumab (Active Comparator): Eligible patients received bevacizumab-EU 15 mg/kg every three weeks for 6 cycles, then 7.5mg/kg until disease progression, intolerable toxicity, withdrawal of consent, lost to follow up or death.
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: TAB008 — 15 mg/kg every three weeks for 6 cycles,then 7.5mg/kg until disease progression, intolerable toxicity, withdrawal of consent, lost to follow up or death
  Arms: TAB008
Drug: Bevacizumab — 15 mg/kg every three weeks for 6 cycles,then 7.5mg/kg until disease progression, intolerable toxicity, withdrawal of consent, lost to follow up or death
  Arms: Bevacizumab

SUMMARY:
In this randomized, double-blind, multicenter, phase III similarity study, treatment naive, EGFR wild-type, locally advanced, metastatic, or recurrent non-squamous, non-small cell, lung cancer (ns-NSCLC) patients were enrolled and randomized (1:1) into TAB008 or Bevacizumab-EU groups. Patients received TAB008 or bevacizumab-EU 15 mg/kg intravenously plus paclitaxel/carboplatin for 4-6 cycles followed by TAB008 or bevacizumab-EU 7.5 mg/kg until disease progression, unacceptable toxicity or death. The primary endpoint compared the objective response rate (ORR) within 6 cycles as read by an independent radiological review committee (IRRC). Secondary endpoints compared disease control rate (DCR) Within 6 cycles, duration of response (DoR), progression free survival (PFS), a year overall survival rate (OSR), overall survival (OS), safety, immunogenicity, and steady state pharmacokinetics.

DETAILED DESCRIPTION:
This randomized, double-blind, equivalence study was conducted in China. Treatment naïve, EGFR wild-type (by PCR or NGS) nsNSCLC patients were enrolled. Patients had to be between 18-75 years of age; stage IIIB to IV pathology confirmed nsNSCLC; ECOG PS 0-1; have adequate organ function; no uncontrollable infectious or serious illnesses; and most importantly, measurable lesion according to Response Evaluation Criteria in Solid Tumor(RECIST) version 1.1. Major exclusion criteria included tumors invading major blood vessels, previous major cardiovascular accidents (stroke, heart attack, uncontrollable hypertension), bleeding diathesis, proteinuria; prior history of malignancy other than NSCLC. Patients underwent tumor assessment using contrast-enhanced CT scans every two cycles for the first six cycles, then every four cycles thereafter until disease progression. Eligible patients were randomized 1:1 to receive TAB008 or bevacizumab-EU 15 mg/kg every three weeks for 6 cycles, then 7.5mg/kg until disease progression, intolerable toxicity, withdrawal of consent, lost to follow up or death. All patients received carboplatin (area under the curve (AUC)=5.0 mg/ml/min) and paclitaxel (175 mg/m2) every three weeks for between 4 to 6 cycles.Eligible subjects were randomized 1:1 by the Interactive Web Response System (IWRS) into the TAB008 group or bevacizumab-EU group.The primary endpoint would be overall response rate (ORR) within the first 6 cycles of treatment determined by the independent radiology review committee (IRRC).

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily participate in the study and sign the informed consent form;
2. Aged 18 to 75 years (inclusive), male or female;
3. Patients with histologically and/or cytologically confirmed, inoperable, locally advanced (Stage IIIb, IIIc), metastatic (Stage IV), or relapsed or progressive non-squamous cell carcinoma after local therapy (in cases of multiple tumor components, the predominant cell type is classified);
4. No sensitive mutation of epidermal growth factor receptor (EGFR) gene (18, 19, 21), no other known activating mutations (such as ALK, ROS) which has treatment approved by NMPA;
5. At least one measurable lesion according to RECIST 1.1 criteria; and this lesion has not received radiotherapy:
6. Definition of measurable disease: Lesions that can be precisely measured in at least one dimension by any of the following: computed tomography (CT) scan or magnetic resonance imaging (MRI) scan with enhanced spiral CT or multidetector CT (MDCT) with extra-nodal lesions at least 10 mm in diameter and lymph node lesions at least 15 mm in short axis when the slice thickness is 5 mm or less；
7. Patients who have never received systemic chemotherapy, anti-angiogenic drug and molecular targeted drug therapy for primary tumor or metastasis (note: subjects who received adjuvant therapy previously are allowed, but only patients who have no progression or recurrence during and within 6 months after completion of adjuvant therapy)；
8. 0 ≤ ECOG PS ≤ 1;
9. Expected survival time ≥ 3 months;
10. The subject has recovered from the damage caused by other local treatments, including radiotherapy or surgery > 4 weeks from the start of study treatment, and the wound has completely healed; however, patients who receive palliative radiotherapy for bone metastases 2 weeks before the start of study treatment can be allowed;
11. Laboratory tests within 14 days before randomization meet the requirements.

Exclusion Criteria:

1. Patients with brain metastases ;
2. History of bleeding diathesis, high risk of bleeding, or coagulopathy, including thrombotic disease within 6 months prior to Screening and/or hemoptysis (≥ 2.5 mL in a single cough) within 3 months prior to Screening;
3. CT/MRI image shows tumor encasement or invasion into the lumen of great vessels (e.g., pulmonary artery or superior vena cava) and patients with bleeding risk judged by the investigator;
4. Uncontrolled hypertension (systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg after combination therapy with two or more antihypertensive agents), and patients with a previous history of hypertensive crisis or hypertensive brain;
5. Significant cardiovascular or cerebrovascular disease;
6. Active peptic ulcer or fracture, active infection at randomization, tracheoesophageal fistula, gastrointestinal perforation or gastrointestinal fistula, and intra-abdominal abscess within 6 months before screening;
7. Patients who have undergone major surgical procedures (including open-heart biopsy), have major trauma, or are expected to require major surgery during the study;
8. Minor surgical procedures (e.g., deep veins, ports) within 24 hours prior to receiving study drug;
9. Moderate to large amount of pericardial effusion, abdominal or pleural effusion that cannot be controlled by pumping or other symptomatic treatment (symptomatic treatment is allowed, but drugs with anti-tumor indications such as chemotherapeutic drugs, anti-angiogenic drugs and molecular targeted drugs cannot be given);
10. Known hypersensitivity to bevacizumab, paclitaxel and carboplatin injection and its excipients;
11. Patients with other malignant tumors except lung cancer within 5 years;
12. Patients who have used other clinical study treatment within 4 weeks before the start of study treatment;
13. History of alcohol or drug abuse;
14. Pregnant and lactating women; women of childbearing potential and male patients who require effective contraceptive methods during the study and for 6 months after administration of study drug;
15. Other conditions that, in the opinion of the investigator, should not be included.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 549 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2020-03-24 (Actual); Study Completion 2020-03-24 (Actual)

PRIMARY OUTCOMES:
ORR | at the end of cycle 6 (each cycle is 21 days).
  The primary endpoint is overall response rate (ORR) within the first 6 cycles of treatment.ORR includes Complete Response Rate and Partial Response Rate.ORR will be independently evaluated by the independent radiology review committee (IRRC).

SECONDARY OUTCOMES:
Disease control rate(DCR) | at the end of cycle 6 (each cycle is 21 days).
  Disease Control Rate is defined as the proportion of patients with complete response(CR), partial response(PR), or stable disease(SD) as defined by RECIST 1.1.
Duration of Response (DoR) | the time from the date of first documented response (CR or PR) until the first date of documented progression or death, and any participant not known to have died at the time of analysis were censored based on the last objective tumor evaluation.
  DoR was defined as the time from the date of first documented response (CR or PR) until the first date of documented progression or death in the absence of disease progression .
PFS | From the date of randomization until the date of objective disease progression or death
  PFS was defined as the time from the date of randomization until the date of objective disease progression or death (by any cause in the absence of progression).
overall survival rate(OSR) at 12 months | 12 months after date of randomization
  12-month OSR was defined as the proportion of patients who have not died at 12 months after randomization over the total number of evaluable patients.
Overall survival(OS) | From the time from the date of randomization until death due to any cause, assessed up to the data cut-off date.
  The OS was defined as the time from the date of randomization until death due to any cause. Any participant not known to have died at the time of analysis were censored based on the last recorded date on which the participant was known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: min liu, doctor, Study Director — No120changyang street ,Suzhou Industrial Park, Jiangsu
Locations (1):
- TOT, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lu S, Qin S, Zhou Z, Chen J, Gu K, Sun P, Pan Y, Yu G, Ma K, Shi J, Sun Y, Yang L, Chen P, Liu A, He J. Bevacizumab biosimilar candidate TAB008 compared to Avastin(R) in patients with locally advanced, metastatic EGFR wild-type non-squamous non-small cell lung cancer: a randomized, double-blind, multicenter study. J Cancer Res Clin Oncol. 2023 Aug;149(9):5907-5914. doi: 10.1007/s00432-022-04563-4. Epub 2023 Jan 3. PMID 36595042